CLINICAL TRIAL: NCT05269173
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase II Clinical Trial to Evaluate the Efficacy and Safety of Flos Gossypii Flavonoids Tablet in the Treatment of Mild and Moderate Alzheimer's Disease
Brief Title: Efficacy and Safety of Flos Gossypii Flavonoids Tablet in the Treatment of Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Xinjiang Uygur Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jianping Jia, Director and Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HJG- MHHZHTP-XJWWEYY
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease
Keywords: medullary sea deficiency; brain collateral stasis syndrome
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active group(low dose group) (Active Comparator): Take 5 tablets each time (including 3 tablets of study drug and 2 tablets of placebo), 3 times a day, a total of 2.7g per day. Take it with warm water half an hour before meals.
  Interventions: Drug: Flos gossypii flavonoids tablet
- Active group(high dose group) (Active Comparator): Take 5 tablets of the study drug each time, 3 times a day, a total of 4.5g per day. Take it with warm water half an hour before meals.
  Interventions: Drug: Flos gossypii flavonoids tablet
- Control group (Placebo Comparator): Take 5 tablets of the control drug (placebo) each time, 3 times a day, 4.5g a day. Take it with warm water half an hour before meals.
  Interventions: Drug: Flos gossypii flavonoids tablet

INTERVENTIONS:
Drug: Flos gossypii flavonoids tablet — The distribution ratio between the groups was 1:1:1, and the stratification factor was the degree of illness CDR score. In the study, the entry of each subject into the high-dose group, low-dose group or placebo group will be determined by the randomized system.

SUMMARY:
In clinical trials of preclinical pharmacodynamic studies, Flos Gossypii Flavonoids Tablet has been proved to significantly improve the learning and memory ability of Alzheimer's disease model. Phase I clinical tolerance test is to observe the human body's tolerance to Flos Gossypii Flavonoids Tablet, and provide a basis for the formulation of safe and reasonable dosing regimens for phase II clinical trials. Therefore, a Phase II clinical trial is now being conducted to explore the efficacy and safety of the Flos Gossypii Flavonoids Tablet in the treatment of mild to moderate Alzheimer's disease (marinus sea deficiency/brain collateral stasis syndrome). In this study, the researchers will use a multicenter, randomized, double-blind, placebo-controlled parallel method to recruit AD patients to confirm the efficacy and safety of Flos Gossypii Flavonoids Tablet. Confirmation of drug efficacy will be observed through changes in AD patients' general cognitive and different cognitive domain functions, daily living activities, and symptom severities.

DETAILED DESCRIPTION:
Cotton flower is a Xinjiang Uygur ethnic medicine, and its main active ingredients are flavonoids. Studies have proved that flavonoids have strong characteristics of antioxidant stress and anti-inflammatory response. Preclinical pharmacodynamic studies on rats showed that the Flos Gossypii Flavonoids Tablet could significantly improve the learning and memory ability of AD model caused by different factors, and the mechanism may be related to its inhibition of oxidative stress and inflammatory response. A total of 57 subjects were enrolled in the Phase I tolerance clinical study. The results showed that the experimental drug may temporarily increase the three indexes of glutamic oxaloacetic transaminase, creatine kinase and lactate dehydrogenase, which can self-recovery in a short time. Combined with the safety evaluation results of phase I clinical trial, Flos Gossypii Flavonoids Tablet is a drug with high safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 to 85 years old (including 50 and 85 years old), male or female;
2. Meet the diagnostic criteria of "likely ad dementia" of the National Institute on aging Alzheimer's disease association (NIA-AA) (2011);
3. The subjects are primary school graduates / graduates and above, and have the ability to complete the cognitive ability test and other tests specified in the program;
4. Memory loss lasted for at least 6 months and tended to worsen gradually;
5. Subjects with mild or moderate illness: 11 ≤ MMSE ≤ 26;
6. Total score of Clinical Dementia Rating Scale (CDR):

   Mild dementia: CDR = 1.0; Moderate dementia: CDR = 2.0;
7. The total score of Hachinski scale(HIS) ≤ 4;
8. The total score of Hamilton Depression Scale (HAMD 17 item version) is ≤ 10;
9. There was no obvious positive sign in nervous system examination;
10. Coronal scanning of head MRI in screening stage: the MTA grade of medial temporal lobe atrophy visual assessment scale is grade 2 or higher, and the signal changes of T2 FLAIR sequence in coronal position of hippocampus. If the subject can provide the head MRI film that meets the requirements within 1 month before screening, it can be used as the basis for enrollment without repeated shooting; If the researcher cannot judge whether the subject's condition has changed, the coronal MRI scan of the head before enrollment can be added;
11. The subjects should have stable and reliable caregivers, who will take care of them at least 3 days a week and at least 2 hours a day. The caregivers will accompany the subjects to participate in the whole process of the study. Caregivers must accompany the subjects to the study visit and assist the investigator in completing the Neuropsychiatric Inventory (NPI), Alzheimer's Disease Collaborative Study-Ability of Daily Living Scale (ADCS-ADL), and Clinician Interview Based Impression of Severity (CIBIC -plus), and other scale scores;
12. Agree to participate and sign the informed consent form by the legal guardian. Due to the subject's limited cognitive ability and other reasons, the subject's signature is allowed to be left blank, and the reason is explained. In addition, the legal guardian shall sign the reason statement, and the legal guardian shall sign the informed consent;
13. Meet the criteria the traditional Chinese medicine of AD which is characterized by the syndrome of insufficient sea of marrow/cerebral collateral stasis. According to the Dementia Syndrome Classification Scale (SDSD), one of the syndromes of insufficient sea of marrow/cerebral collateral stasis can be met.

Exclusion Criteria:

1. During screening, MRI examination showed significant focal lesions, fulfilling one of the following conditions:

   ① There were more than 2 infarcts with diameter > 2 cm at any site;

   ② MRI examination showed that there were infarcts with arbitrary diameter in key parts (such as thalamus, hippocampus, entorhinal cortex, paraolfactory cortex, angular gyrus, cortex and other subcortical gray matter nuclei);

   ③ Fazekas scale grade of white matter lesions > 2;

   ④ There are other imaging evidences that do not support mild and moderate AD;
2. Dementia caused by other reasons: vascular dementia, central nervous system infection, Creutzfeldt Jakob disease, Huntington's disease, Parkinson's disease, Lewy body dementia, traumatic dementia, other physical and chemical factors (such as drug poisoning, alcoholism, carbon monoxide poisoning, etc.), important physical diseases (such as hepatic encephalopathy, pulmonary encephalopathy, etc.), intracranial space occupying lesions (such as subdural hematoma, brain tumor), endocrine disorders (such as thyroid disease, parathyroid disease), and vitamin B12, folic acid deficiency or any other known cause;
3. Have suffered from central nervous system diseases (including stroke, optic neuromyelitis, epilepsy, etc.);
4. Subjects who were diagnosed with psychiatric disorders according to DSM-V criteria, including schizophrenia or other mental diseases, bipolar disorder, severe depression or delirium;
5. Abnormal laboratory indexes: liver function (ALT and AST) exceeded 1.5×ULN, renal function (CR) exceeded 1.5×ULN, and creatine kinase exceeded 2×ULN;
6. Untreated hypertensive and hypotensive subjects at screening, or hypertensive subjects with uncontrolled hypertension after treatment; subjects with good blood pressure control after treatment can be determined by the investigator to be suitable for inclusion in this study;
7. Within 1 month of the screening visit, the subject has new or ongoing unstable or serious heart, lung, liver, kidney and hematopoietic diseases according to the judgment of the researcher, and does not meet the conditions for clinical research;
8. Clinically, people with significant allergic reaction history, especially drug allergy history, or known allergy to this product and its excipients;
9. Dyspepsia, esophageal reflux, gastric bleeding or peptic ulcer disease, frequent heartburn (≥ once a week) or any surgical operation that may affect drug absorption (such as partial / total gastrectomy, partial / total small bowel resection and cholecystectomy) within 6 months before screening;
10. Alcohol or drug abusers;
11. Human immunodeficiency virus antibody (ant HIV) and Treponema pallidum antibody (ant TP) are positive;
12. Those who are currently using and cannot stop using drugs for Alzheimer's disease;
13. Screening for cholinesterase inhibitors, N-methyl-D-aspartate receptor antagonists (NMDA antagonists), mental retardants, antiparkinsonian drugs and opioid analgesics taken within 1 month before the visit;
14. There are uncorrectable visual and auditory disorders, and the neuropsychological test and scale evaluation cannot be completed;
15. Female subjects with positive pregnancy test or lactation and subjects unable to take effective contraceptive measures or have family planning;
16. Participated in other clinical trials within 3 months before the screening visit;
17. There are other situations that the researcher believes are not suitable to participate in this study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive section(ADAS-cog/11) | Change from baseline in ADAS-cog scores at Week 26
  Differences between the low-dose and high-dose groups in changes in ADAS cog/11 scores (relative to baseline) at weeks 13 and 26 were compared with the placebo group.
  The ADAS-cog/11 measures 11 items: word recall, commands, constructional praxis, naming objects or fingers, ideational praxis, orientation, word recognition, remembering word recognition test instructions, spoken language ability, word-finding difficulty and comprehension. The total score ranges from 0 to 70, with lower scores representing milder disease.

SECONDARY OUTCOMES:
Mini-mental State Examination (MMSE) | Change from baseline in MMSE scores at Week 26
  Differences between the low-dose and high-dose groups in changes in MMSE scores (relative to baseline) at weeks 13 and 26 were compared with the placebo group.
  The MMSE scale can reflect the mental state and the degree of cognitive impairment of the subjects, with a total score of 30 points. The higher the score, the better the subject's condition.
Alzheimer's Disease Co-operative Study Activities of Daily Living (ADCS-ADL) | Change from baseline in ADCS-ADL scores at Week 26
  Differences between the low-dose and high-dose groups in changes in ADCS-ADL scores (relative to baseline) at weeks 13 and 26 were compared with the placebo group.
  The ADCS-ADL scale can reflect the degree of impairment of the subjects' daily life ability, with a total score of 78 points. The higher the score, the better the subjects' living ability.
Clinician Interview Based Impression of Severity (CIBIC-plus) | Change from baseline in CIBIC-plus scores at Week 26
  Differences between the low-dose and high-dose groups in changes in CIBIC-plus scores (relative to baseline) at weeks 13 and 26 were compared with the placebo group.
  The CIBIC-plus scale is based on interviews with patients and their caregivers by research physicians to ask, record and assess changes in patients' conditions. Outcomes assessed were: Caregiver Meeting-Clinical Impression Change, Subject Meeting-Clinical Impression Change, and Overall Clinical Impression Change.
Neuropsychiatric Inventory (NPI) | Change from baseline the scores of 12 behavioral domains in NPI at Week 26.
  Differences in changes in 12-item behavioral domain scores (relative to baseline) on the NPI scale at weeks 13 and 26 between the low-dose and high-dose groups compared with placebo.
  The NPI scale is an interview conducted by the research doctor based on the patient's caregiver to ask the patient's mental and emotional changes. The questions included 12 items including delusions, hallucinations, depression, and anxiety, each of which identified the severity, frequency, and psychological stress of the caregiver.
Neuropsychiatric Inventory (NPI) | Change from baseline in Caregiver Stress Score on the NPI Scale at Week 26
  Differences in changes in caregiver stress scores (relative to baseline) on the NPI scale at weeks 13 and 26 between the low-dose and high-dose groups compared with placebo.
Dementia syndrome classification scale (SDSD) | Change from baseline in SDSD scores at Week 26
  Differences between the low-dose and high-dose groups in changes in SDSD scores (relative to baseline) at week 26 were compared with the placebo group.
  This project selects the type of medullary sea insufficiency and the type of brain collateral stasis from the SDSD scale for evaluation. The maximum score for the assessment is 30 points. If the total score is less than 7 points, the syndrome is not established, and if the total score is ≥ 7 points, the syndrome is established.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Hefei Second People's Hospital, Hefei, Anhui
  - Lu'an Hospital of traditional Chinese Medicine, Lu'an, Anhui
  - Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Oriental Hospital of Beijing University of traditional Chinese Medicine, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Sun Yat Sen Memorial Hospital of Sun Yat sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - Daqing People's Hospital, Daqing, Heilongjiang
  - Luoyang First Hospital of traditional Chinese Medicine, Luoyang, Henan
  - Jiangsu Hospital of traditional Chinese Medicine, Nanyang, Jiangsu
  - Taizhou Hospital of traditional Chinese Medicine, Taizhou, Jiangsu
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu
  - PLA Northern Theater Air Force Hospital, Shenyang, Liaoning
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Hospital of traditional Chinese Medicine, Xi’an, Shanxi
  - Xi'an High Tech Hospital, Xi’an, Shanxi
  - Xidian Group Hospital, Xi’an, Shanxi
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: No